CLINICAL TRIAL: NCT01466621
Title: Response to Cardiac Resynchronization Therapy of Previously Right Ventricular Paced Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ISRCRM110009(Boston Sci Corp)
Record Dates: First submitted 2011-11-02; First posted 2011-11-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure; Pacing Induced Dyssynchrony
Keywords: cardiac resynchronization therapy; heart failure; mortality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Previously RV Paced: Patients who were RV paced prior to receiving a cardiac resynchronization therapy device.
- Non-Previously RV Paced: Patients who received a CRT device without being previously RV paced.

SUMMARY:
The present proposal is designed to investigate the response to CRT in patients who were previously paced from the right ventricle (RV). The negative physiologic and structural changes associated with chronic RV pacing are well documented, but patient response following upgrade to CRT after chronic RV pacing has not been well characterized in a large cohort.

DETAILED DESCRIPTION:
The RV apex has historically been used as the site for ventricular pacing in cases of sinus node dysfunction or atrioventricular block because of its relatively accessible location for lead implantation. Initial studies showed RV pacing improved symptoms, exercise capacity, quality of life, and survival in these patients.11-13 However, more recent studies have illustrated that chronic RV pacing may actually impair LV systolic function and increase the risks of heart failure, hospitalization, and death in some patients.

The primary hypothesis is that patients upgraded to CRT from a RV pacemaker respond better than those receiving CRT as a first time device. To test this hypothesis the investigators will compare changes in cardiac size and function, and hospitalization and survival rates between the two patient groups.

The second hypothesis will investigate whether changes in septal dyssynchrony are correlated with changes in ejection fraction in previously RV paced patients. The investigators believe that the patients with the most improvement in septal dyssynchrony due to RV pacing will see the greatest improvement in LV function following upgrade to CRT. A significant correlation between change in IM-S and change in EF will support the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Received a CRT device between 2003 and 2009 at United Heart & Vascular Clinic
* QRS duration > 120 msec
* Pre-CRT ejection fraction =< 35%

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective review of patients receiving CRT at United Heart & Vascular Clinic between 2003 and 2009.
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Death from any cause | Average of 4 years
  Retrospectively measure the time in days from device implant to death, if applicable.
Cardiovascular Hospitalization | Average of 4 years
  Retrospectively measure the time in days from device implant to hospitalization, if applicable.

SECONDARY OUTCOMES:
Change in ejection fraction | Approximately one year
  A measure of cardiac performance.

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, MD, Principal Investigator — United Heart & Vascular Clinic
Locations (1):
- United Heart & Vascular Clinic, Saint Paul, Minnesota, United States